CLINICAL TRIAL: NCT07037940
Title: Comparing Clinical Key AI and GPT-4 for Diagnostic Reasoning and Management Decisions
Brief Title: Physician Response Evaluation With Contextual Insights vs. Standard Engines - Artificial Intelligence RAG vs LLM Clinical Decision Support
Acronym: PRECISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-16599
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Large Language Models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OpenEvidence (Active Comparator): Participants in this arm will use OpenEvidence as their research tool
  Interventions: Other: OpenEvidence
- ChatGPT (Active Comparator): Patients in this arm will use Chat-GPT as their research tool
  Interventions: Other: GPT-4

INTERVENTIONS:
Other: OpenEvidence — Medical information platform which uses retrieval-augmented generation to access medical literature
  Arms: OpenEvidence
Other: GPT-4 — A chatbot application developed that uses GPT-4, a large language model, to engage in conversational interactions with users.
  Other Names: ChatGPT
  Arms: ChatGPT

SUMMARY:
Clinical decision support tools powered by artificial intelligence are being rapidly integrated into medical practice. Two leading systems currently available to clinicians are OpenEvidence, which uses retrieval-augmented generation to access medical literature, and GPT-4, a large language model. While both tools show promise, their relative effectiveness in supporting clinical decision-making has not been directly compared. This study aims to evaluate how these tools influence diagnostic reasoning and management decisions among internal medicine physicians.

DETAILED DESCRIPTION:
Internal medicine attendings and residents are invited to participate in a study investigating how physicians using a RAG-based LLM (OpenEvidence) perform compared to those using a standard general-purpose LLM (ChatGPT) on both diagnostic reasoning and complex management decisions. As AI tools increasingly enter clinical practice, evidence is needed about which approaches best support physician decision-making. This study will help determine if specialized medical knowledge retrieval systems (OpenEvidence) provide advantages over general AI assistants (ChatGPT) when solving real clinical cases.

Participants will complete one 90-minute Zoom session where clinical cases derived from real, de-identified patient encounters will be solved. Participants will be randomly assigned to use either OpenEvidence or ChatGPT and all responses evaluated by blinded scorers using a validated rubric.

Note that this exempted study will compare OpenEvidence (as opposed to Clinical Key AI) vs ChatGPT although the official study title suggests otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residents
* Internal medicine attending physicians

Exclusion Criteria:

* Not meeting Inclusion Criteria

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Reasoning Performance as determined by Rater Scores | 15-minutes upon completion of cases, up to approximately 90 minutes total
  Clinical reasoning performance will be evaluated based upon the accuracy of the rater scores to responses to the surveys administered. Six blinded, trained independent raters will independently score each participant's response using a validated scoring rubric. Possible response scores can range from 0-100% with higher scores indicating increased clinical reasoning performance. Results for each assessment will be summarized by study arm using basic descriptive statistics and analyzed using mixed-effects models to account for within-subject correlation and between-subject factors.

SECONDARY OUTCOMES:
Time efficiency | Up to approximately 75 minutes
  Time efficiency will be assessed based on the amount of time it takes for participants to complete the surveys. Each survey will automatically be time stamped to record the amount of time needed for each participant to answer each case. Results for the virtual session will be summarized by study arm using basic descriptive statistics and analyzed.
Decision confidence | 15-minutes upon completion of cases, up to approximately 90 minutes total
  Decision confidence will be determined by asking participants to assess the level of confidence in survey answers using a scale ranging from 1-5 (1 being least confident, 5 being most confident) such that higher scores are associated with increased confidence in responses. Scores will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Shitij Arora, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Harvard Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - MontefioreMC, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabral S, Restrepo D, Kanjee Z, Wilson P, Crowe B, Abdulnour RE, Rodman A. Clinical Reasoning of a Generative Artificial Intelligence Model Compared With Physicians. JAMA Intern Med. 2024 May 1;184(5):581-583. doi: 10.1001/jamainternmed.2024.0295. PMID 38557971
- [Background] Singhal K, Azizi S, Tu T, Mahdavi SS, Wei J, Chung HW, Scales N, Tanwani A, Cole-Lewis H, Pfohl S, Payne P, Seneviratne M, Gamble P, Kelly C, Babiker A, Scharli N, Chowdhery A, Mansfield P, Demner-Fushman D, Aguera Y Arcas B, Webster D, Corrado GS, Matias Y, Chou K, Gottweis J, Tomasev N, Liu Y, Rajkomar A, Barral J, Semturs C, Karthikesalingam A, Natarajan V. Large language models encode clinical knowledge. Nature. 2023 Aug;620(7972):172-180. doi: 10.1038/s41586-023-06291-2. Epub 2023 Jul 12. PMID 37438534
- [Background] Strong E, DiGiammarino A, Weng Y, Kumar A, Hosamani P, Hom J, Chen JH. Chatbot vs Medical Student Performance on Free-Response Clinical Reasoning Examinations. JAMA Intern Med. 2023 Sep 1;183(9):1028-1030. doi: 10.1001/jamainternmed.2023.2909. PMID 37459090
- [Background] Schaye V, Miller L, Kudlowitz D, Chun J, Burk-Rafel J, Cocks P, Guzman B, Aphinyanaphongs Y, Marin M. Development of a Clinical Reasoning Documentation Assessment Tool for Resident and Fellow Admission Notes: a Shared Mental Model for Feedback. J Gen Intern Med. 2022 Feb;37(3):507-512. doi: 10.1007/s11606-021-06805-6. Epub 2021 May 4. PMID 33945113
- [Background] Goh E, Gallo R, Hom J, Strong E, Weng Y, Kerman H, Cool JA, Kanjee Z, Parsons AS, Ahuja N, Horvitz E, Yang D, Milstein A, Olson APJ, Rodman A, Chen JH. Large Language Model Influence on Diagnostic Reasoning: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2440969. doi: 10.1001/jamanetworkopen.2024.40969. PMID 39466245
- [Background] Goh E, Gallo RJ, Strong E, Weng Y, Kerman H, Freed JA, Cool JA, Kanjee Z, Lane KP, Parsons AS, Ahuja N, Horvitz E, Yang D, Milstein A, Olson APJ, Hom J, Chen JH, Rodman A. GPT-4 assistance for improvement of physician performance on patient care tasks: a randomized controlled trial. Nat Med. 2025 Apr;31(4):1233-1238. doi: 10.1038/s41591-024-03456-y. Epub 2025 Feb 5. PMID 39910272